CLINICAL TRIAL: NCT06256939
Title: Therapy BRIDGE (Bringing Real-Time Instruction Via Developmental and Gestationally-appropriate Education/Coaching) Program: A Pilot Study
Acronym: Therapy BRIDGE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Responsible Party: Principal Investigator, Grace Sagester, Co-Principal Investigator, Occupational Therapist, Division of Occupational & Physical Therapy, Children's Hospital Medical Center, Cincinnati
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2023-0236
Record Dates: First submitted 2024-01-04; First posted 2024-02-13 (Actual); Last update posted 2025-02-20 (Actual); Status verified 2025-02

CONDITIONS: Intraventricular Hemorrhage
Keywords: IVH; NICU; caregiver education; occupational therapy; physical therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention Group (Experimental): The Therapy BRIDGE program is a prospective, longitudinal, non-randomized pilot study for infants diagnosed with IVH and their caregivers. The Therapy BRIDGE program will begin as the infant is nearing discharge from the NICU and continue as the infant transitions to home. It will use a hybrid model including both in-person and telehealth sessions.
  Interventions: Other: Therapy BRIDGE Program
- Control Group (No Intervention): In the instance that a patient is deemed eligible to participate in the Therapy BRIDGE program and the caregiver chooses not to participate, the caregiver will be offered the opportunity to be enrolled in the control arm of our study as part of a monitoring group. This group of patients will continue to receive usual care while admitted to the NICU and any outpatient recommendations will be deferred to the primary NICU therapists caring for the infant based on the patient's individualized needs.

INTERVENTIONS:
Other: Therapy BRIDGE Program — A standardized education and coaching intervention will be developed to promote optimal neurodevelopmental outcomes through caregiver empowerment. This pilot study will enroll up to 15 infants with IVH and their caregivers during their NICU stay. These infant-caregiver dyads will receive up to 10 sessions utilizing the Therapy BRIDGE program over a four-month period that spans the hospital to home transition.
  Arms: Intervention Group

SUMMARY:
The goal of this pilot study is to develop a novel caregiver education and coaching intervention for infants with intraventricular hemorrhage (IVH) and their caregivers during the NICU to home transition. The main questions it aims to answer are:

1. Development of a novel caregiver education and coaching intervention focused on infant development and caregiver needs to "bridge the gap" during the NICU to home transition
2. Pilot test the feasibility, acceptability, and efficacy of this program for infants with intraventricular hemorrhage (IVH) and their caregivers.

DETAILED DESCRIPTION:
Infants born preterm are often medically complex and at high-risk for neurodevelopmental challenges. During their Neonatal Intensive Care Unit (NICU) stay, infants and caregivers receive continuous support and have constant access to a variety of specialists. Research has shown that caregiver involvement in their infant's care in the NICU helps to improve outcomes. However, caring for these infants upon discharge can be overwhelming to caregivers. Currently, there is no formal intervention in place to support caregivers as they transition their infant home. The overall objectives of the Therapy BRIDGE program are to (1) create a novel caregiver education and coaching intervention focused on infant development and caregiver needs to "bridge the gap" during the NICU to home transition and (2) pilot test the feasibility, acceptability, and efficacy of this program for infants with intraventricular hemorrhage (IVH) and their caregivers.

A standardized education and coaching intervention will be developed to promote optimal neurodevelopmental outcomes through caregiver empowerment. This pilot study will enroll up to 15 infants with IVH and their caregivers during their NICU stay. These infant-caregiver dyads will receive up to 10 sessions utilizing the Therapy BRIDGE program over a four-month period that spans the hospital to home transition. Feasibility and acceptability will be measured with caregiver and therapist questionnaires using a 5-point Likert Scale. Intervention efficacy will be measured by administering the Canadian Occupational Performance Measure (COPM) before and after completion of the program and evaluating change scores.

ELIGIBILITY:
Inclusion Criteria for infant participants:

* A diagnosis of IVH, regardless of age at time of enrollment
* Admission to the Cincinnati Children's Hospital NICU

Inclusion Criteria for caregiver participants:

* Must be at least 18 years of age
* Can provide written consent
* Able to participate in the sessions and data collection process

Exclusion Criteria for infant and caregiver participants:

* Transfer out of the NICU prior to discharge or require tracheostomy with ventilator dependence as they will not be discharged directly from the CCHMC NICU
* Infants and caregivers who live outside of the CCHMC service area and will not be eligible for follow up with CCHMC therapies will be excluded.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2023-11-16 (Actual); Primary Completion 2024-09-30 (Actual); Study Completion 2024-09-30 (Actual)

PRIMARY OUTCOMES:
Canadian Occupational Performance Measure (COPM) | At enrollment and through study completion, an average of 2 months
  A client-centered outcome measure that helps identify and prioritize barriers that limit participation in meaningful activities (e.g., play, feeding, sleep, etc.). The COPM is a valid, responsive, and reliable scale that allows researchers to determine clinically significant changes in participants' performance and satisfaction. Participants will rate items on a scale of 1-10 with the average performance/satisfaction scores calculated (higher correlates with higher satisfaction/performance).

SECONDARY OUTCOMES:
Caregiver Questionnaire of Perceived Feasibility & Acceptability of Therapy BRIDGE Program | At enrollment and through study completion, an average of 2 months
  Caregiver questionnaire to measure feasibility and acceptability. Participants will rate items on a scale of 1-5 with the average scores calculated (higher correlates with higher acceptance/performance).
Therapist Questionnaire of Acceptability of Therapy BRIDGE Program | To be completed at study completion, an average of 2 months after enrollment
  Questionnaire to measure therapist's acceptability of novel education program. Participants will rate items on a scale of 1-5 with the average scores calculated (higher correlates with higher acceptance/performance).

CONTACTS AND LOCATIONS:
Overall Officials: Grace Sagester, OTD, OTR/L, BCP, Principal Investigator — Children's Hospital Medical Center, Cincinnati; Ashley Pinger, PT, DPT, PCS, Principal Investigator — Children's Hospital Medical Center, Cincinnati
Locations (1):
- Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio, United States

IPD SHARING:
Plan to Share IPD: No